CLINICAL TRIAL: NCT06540703
Title: Ketogenic Diet in Weight Recovered Anorexia Nervosa to Normalize Brain Metabolism and Persistent Eating Disorder Psychopathology
Brief Title: Ketogenic Diet and Brain Response in Anorexia Nervosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810326
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: therapeutic ketogenic diet for 14 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Ketogenic Diet (Experimental): Subjects will be placed on a therapeutic ketogenic diet (TKD) for a duration of 14 weeks.
  Interventions: Dietary Supplement: Therapeutic Ketogenic Diet (TKD)

INTERVENTIONS:
Dietary Supplement: Therapeutic Ketogenic Diet (TKD) — 2 week induction to establish ketosis followed by 12 weeks therapeutic ketogenic diet

SUMMARY:
This is a longitudinal study with an open design in weight recovered anorexia nervosa (wrAN) individuals. Healthy controls (HC) will also be assessed. Study participants will be carefully assessed and will have 18F-fluorodeoxyglucose ([18F]FDG) positron emission tomography (PET) scans for assessment of regional brain glucose uptake. The wrAN group will be compared to healthy controls. Participants in the wrAN group will then complete 14 weeks of therapeutic ketogenic diet (TKD). At the end of the TKD study, participants will have assessments and a second [18F]FDG and TMS/EEG scan. Study participants will be followed over six months after the intervention. This follow-up procedure will help determine whether symptom improvement will be stable or worsen in individuals who choose to continue or discontinue the TKD intervention. This will be a naturalistic follow-up.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a severe psychiatric disorder. However, neurobiological models and interventions to explain and treat the core characteristics of food restriction, feeling fat, and body size overestimation are lacking. While research has made progress in understanding brain function involved in AN pathophysiology, translating those results into biological therapies has been challenging. Studies have suggested that metabolic factors contribute to developing and maintaining AN pathophysiology. Specifically, brain glucose utilization and metabolism may be altered in AN, interfere with brain energy homeostasis, and contribute to illness development and maintenance. A small study indicated that ketosis might be therapeutic for AN core behaviors such as eating and shape concerns. In this application, the investigator will study individuals weight recovered from AN, establish biological targets as diet-related metabolic markers for AN (R61 phase), and replicate and link those targets to AN-specific behaviors (R33 phase). The weight recovered AN group will also be compared with a healthy control sample. The R61 Phase Specific Aim of the project is to establish target engagement for a therapeutic ketogenic diet (TKD) in AN after weight recovery and establish safety and tolerability. It is hypothesized that TKD will be associated with reduced brain glucose metabolism using [18F]fluorodeoxyglucose ([18F]FDG) and positron emission tomography (PET) (target engagement). Higher blood ketosis levels will be associated with a more significant reduction of the brain [18F]FDG glucose metabolism rate (dose dependency). It is hypothesized that TKD will be well tolerated, that participants will remain within the normal weight range (tolerability), and that study participants will be able to adhere to TKD as indicated by regular blood ketosis measurements (treatment fidelity). There will be an initial indication that TKD and associated biological measures correlate with behavioral measures derived from eating disorder-specific assessments.

ELIGIBILITY:
Inclusion Criteria:

Weight Recovered Anorexia Nervosa (wrAN)

* Age 18-45 years old
* Male and Female sexes
* All ethnic backgrounds
* History of restricting-type anorexia nervosa (AN) according to DSM-5 criteria
* Weight recovered with a body mass index > 17.5 for at least one month at the time of study
* Elevated eating disorder-relevant behaviors on the Eating Disorders Inventory-3 and the Eating Disorder Examination Questionnaire

Healthy Control Group

* Age 18-45 years old
* Male and Female sexes
* All ethnic backgrounds
* Normal lifetime BMI according to CDC

Exclusion Criteria:

Weight Recovered Anorexia Nervosa (AN)

* Current pregnancy or nursing (will have to agree to contraceptive measures if sexually active)
* Lifetime history of bipolar I disorder or psychosis
* Current substance abuse or dependence in the past 3 months
* Psychotic illness/other organic brain syndromes, dementia, somatization disorders or conversion disorders
* History of significant head trauma
* Indication of intellectual disability or autism spectrum disorder

Healthy Control Group

* No lifetime psychiatric illness and in particular no eating disorder history
* Not be taking medication, and will not have a first degree relative with an eating disorder.

No subject in either group will have or be

* mental retardation or pervasive developmental disorder
* organic brain syndrome
* dementia
* psychotic disorder
* bipolar disorder
* somatic symptom
* conversion disorder
* current alcohol or substance use disorder
* indication of major medical illness including a history of seizure disorder
* pregnant or nursing at the time of the study
* a history of traumatic brain injury.
* diabetes mellitus or other metabolic disorders that could worsen on a ketogenic diet
* intracranial or any other metal object within or near the head that cannot be safely removed, excluding the mouth
* implanted neurostimulators, intracardiac lines, or heart disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
[18F]fluorodeoxyglucose (FDG) uptake | Difference in pre/post Therapeutic Ketogenic Diet PET/CT scans
  To test whether TKD will be associated with reduced brain [18F]fluorodeoxyglucose (FDG) uptake

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States